CLINICAL TRIAL: NCT01522378
Title: Cardiac Resynchronization and MIBG Imaging
Brief Title: Cardiac Resynchronization and Iodine Meta-Iodobenzylguanidine (MIBG) Imaging
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated because the funding was withdrawn.
Sponsor: Mayo Clinic (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Yong-Mei Cha, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-006296
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Congestive Heart Failure
Keywords: cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Biv-ICD (Experimental): Subjects will be imaged with 123 iodine metaiodobenzylguanidine.
  Interventions: Drug: 123 iodine metaiodobenzylguanidine

INTERVENTIONS:
Drug: 123 iodine metaiodobenzylguanidine — 10 millicurie (mCi) (370 MBq)
  Other Names: AdreView

SUMMARY:
Subjects were recruited if their healthcare provider decided that they needed treatment with a special Internal Cardiac Defibrillator (ICD) called a biventricular ICD. The investigators did this study to see if part of the nerve organ, called the sympathetic nervous system, may be responsible for the improvement seen in patients that receive biventricular pacing. The investigators had three ways to measure sympathetic nervous activity: 1) by using a special blood sample, 2) by monitoring heart rhythm, and 3) by performing a special heart scan.

DETAILED DESCRIPTION:
The Specific Aim #1 of this study is to assess, with 123iodine metaiodobenzylguanidine (123I-MIBG imaging), whether cardiac resynchronization therapy (CRT) rebalances and improves the integrity and function of sympathetic nerve terminals in the failing myocardium. The study will test the hypothesis that resynchronization of biventricular contractility attenuates excessive sympathetic drive, and improves autonomic function and cardiac performance.

The Specific Aim #2 of this study is to determine the relationship between 123I-MIBG labeling of sympathetic activity and physiological measures of cardiopulmonary and autonomic function. This aim is to test the hypothesis that impaired cardiac sympathetic activity, determined by 123I-MIBG imaging will be associated with poorer submaximal exercise gas exchange (higher ventilation - carbon dioxide (CO2) slopes, low end tidal CO2, reduced oxygen pulse and a more rapid frequency response) as well as reduced heart rate power spectral frequencies, a blunted response to positional changes and a delayed heart rate recovery.

ELIGIBILITY:
Inclusion criteria: Indications for Biv-ICD implantation

1. Chronic moderate to severe congestive heart failure (CHF) (NYHA class II or IV)
2. Left ventricular ejection fraction (LVEF) of 35% or less
3. Q wave, R wave and S wave (QRS complex) QRS duration of 120 ms or more
4. On optimized anti-heart failure medical regimen
5. Meet one of the following indications for ICD

   * Survivors of cardiac arrest due to ventricular fibrillation (VF) or ventricular tachycardia (VT) or spontaneous sustained VT
   * Nonsustained VT with coronary disease, prior myocardial infarction, LVEF 35% or less, and inducible VF or sustained VT at electrophysiologic study
   * LVEF of 30% or less with severe coronary artery disease

Exclusion criteria:

1. Patient condition is unstable
2. Patient is unable to give informed consent
3. Not feasible for patient to be followed at Mayo Clinic
4. Female in pregnancy and breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in 123I-MIBG parameters | baseline, 6 months
  changes in 123I-MIBG parameters with cardiac performance including LVEF, stroke volume (SV), left ventricle (LV) and left atrium (LA) dimension, distance of 6-minute walk, NYHA class, and ventricular arrhythmic burden

SECONDARY OUTCOMES:
Change in submaximal exercise gas exchange | baseline, 6 months
  Subjects will perform simplified low intensity cardiopulmonary exercise testing in our laboratory where they breathe for 1 min at rest, perform graded step exercise, increasing from 60, 90, 120 steps per minute until achieving a perceived exertion of 12-14 on the 6-20 Borg scale. This will be followed by a 1 min recovery. Subjects will be instrumented with ECG, pulse oximeter and breathe on a mouthpiece where ventilation, oxygen and carbon dioxide are measured continuously to calculate the desired parameters of ventilatory efficiency (VE/VCO2), PetCO2 and oxygen pulse (O2Pulse) on a breath by breath basis.
Change in Autonomic function | baseline, 6 months
  In addition to the simplified submaximal step test, subjects will also perform a simplified battery of tests for autonomic function. This will include supine to upright measures of heart rate and heart rate variability (HRV), paced breathing (slow to faster frequencies) as well as tracking HRV and responses to the increased metabolic demands of exercise and into recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Cha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No